CLINICAL TRIAL: NCT00339326
Title: Cofactors for Classical Kaposi's Sarcoma and for Kaposi's Sarcoma-Associated Herpesvirus Infection: A Case-Control Study in Sicily
Brief Title: Risk Factors for Non-HIV-Related Kaposi s Sarcoma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902282; 02-C-N282
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2020-05

CONDITIONS: Kaposi's Sarcoma
Keywords: Human Herpes virus 8 (HHV8); Kaposis sarcoma (KS); Kaposi Sarcoma; Karposi Sarcoma-Associated Herpesvirus; KSHV; KS
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (2):
- Cases with Kaposi's Sarcoma: Cases with Kaposi's Sarcoma from Southern Italy.
- Controls without KS: Controls from Southern Italy.

SUMMARY:
This study will try to identify risk factors for Kaposi s sarcoma, a rare skin cancer, and to understand the role of the KSHV virus in development of the disease.

All native-born Italians 21 years of age or older residing in Sicily from July 1, 2002 through June 30, 2005 who have Kaposi s sarcoma not related to HIV infection may be eligible for this study. Healthy control subjects will also be enrolled.

All participants will be interviewed about their childhood, jobs, habits, medical conditions, and treatments. They also will provide a blood sample and a saliva sample, obtained by swishing a mouthwash for 45 seconds and spitting it into a container.

Blood will be tested for two viruses KSHV and HIV that are related to Kapsosi s sarcoma. The KSHV virus is newly discovered and not well understood. In general, a positive KSHV test probably means an infection with the virus has occurred in the past, but not necessarily that disease has developed. HIV is the virus that causes AIDS. People with AIDS have a high risk of Kapsosi s sarcoma. Although HIV and AIDS are very rare among older adults in Sicily, the presence of HIV must be ruled out in order to understand how KSHV is related to Kapsosi s sarcoma.

The blood may also be used to measure immunity (the body s defense against infection and cancer) and for genetic studies to help discover why Kapsosi s sarcoma occurs.

DETAILED DESCRIPTION:
Persons infected with the Kaposi s sarcoma-associated herpesvirus (KSHV) are at risk for developing Kaposi s sarcoma (KS), but the risk factors for KSHV infection and for KS following infection are not well defined. Classical KS (cKS) occurs without apparent immune deficiency (such as AIDS or an allograft). The proposed study will test specific hypotheses and generate new hypotheses on the risk of cKS among persons who have antibodies against KSHV, on the risk of KSHV seropositivity, and on the risk of active KSHV infection, defined as KSHV viremia or viral shedding in saliva. To do so, 120 incident cases of cKS from throughout Sicily and approximately 1800 persons (15% KSHV seropositive) of similar age, sex, and community size will be asked to participate by providing questionnaire data and blood and saliva specimens. Residual formalin-fixed, paraffin embedded tissue from KS skin biopsies will be available for verification of diagnosis and molecular analyses. Primary hypotheses are focused on host genetic susceptibility, endogenous clinical conditions (such as asthma and allergy), and exogenous exposures (cigarette smoking and contact with certain plants, water and soil) that are postulated to affect KSHV activation, dissemination, and disease induction. The study will have sufficient statistical power to detect factors that increase the risk of KSHV seropositivity by 1.5- to 2-fold, the risk of cKS by 2- to 3-fold, and the risk of KSHV viremia or shedding by 3- to 4-fold.

ELIGIBILITY:
* INCLUSION CRITERIA - CASES:

All non-AIDS, pathologically confirmed cases of KS (International Classification of Diseases for Oncology code M9140/3) in native born Italians resident in Sicily from 01 July 2002 through 30 June 2005 (3 years).

EXCLUSION CRITERIA - CASES:

AIDS, history of organ transplant, no pathologic confirmation, not born in Italy, not resident in Sicily, unable to provide informed consent, age less than 21.

INCLUSION CRITERIA - CONTROLS:

Native born Italians, resident in Sicily, on the GP's roster.

EXCLUSION CRITERIA - CONTROLS:

AIDS, history of KS, spouse or relative of an enrolled KS case or of another control, history of organ transplant, not born in Italy, not resident in Sicily, unable to provide informed consent, age less than 21.

Exclusion of children.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population based samples of adults from Italy (Southern Italy).@@@
Sampling Method: Probability Sample
Enrollment: 1383 (Actual)
Dates: Start 2002-09-01; Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Kaposi sarcoma (KS) | 5 years
  Kaposi sarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Sam M Mbulaiteye, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Universita Degli Studi Di Palermo, Palermo, Italy

REFERENCES:
- [Background] Cottoni F, Masala MV, Budroni M, Rosella M, Satta R, Locatelli F, Montesu MA, De Marco R. The role of occupation and a past history of malaria in the etiology of classic Kaposi's sarcoma: a case-control study in north-east Sardinia. Br J Cancer. 1997;76(11):1518-20. doi: 10.1038/bjc.1997.587. PMID 9400951
- [Background] Touloumi G, Hatzakis A, Potouridou I, Milona I, Strarigos J, Katsambas A, Giraldo G, Beth-Giraldo E, Biggar RJ, Mueller N, Trichopoulos D. The role of immunosuppression and immune-activation in classic Kaposi's sarcoma. Int J Cancer. 1999 Sep 9;82(6):817-21. doi: 10.1002/(sici)1097-0215(19990909)82:63.0.co;2-7. PMID 10446447
- [Background] Ziegler JL, Newton R, Katongole-Mbidde E, Mbulataiye S, De Cock K, Wabinga H, Mugerwa J, Katabira E, Jaffe H, Parkin DM, Reeves G, Weiss R, Beral V. Risk factors for Kaposi's sarcoma in HIV-positive subjects in Uganda. AIDS. 1997 Nov;11(13):1619-26. doi: 10.1097/00002030-199713000-00011. PMID 9365767